CLINICAL TRIAL: NCT06114095
Title: Single Cell Sequencing and Multidimensional Omics Studies in Cardiovascular and Neurological Diseases
Status: Recruiting | Type: Observational
Sponsor: Tao Xin (Other)
Responsible Party: Sponsor-Investigator, Tao Xin, Director of Neurosurgery, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(038)
Record Dates: First submitted 2023-10-19; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Nervous System Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Nervous System Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease group: Disease-specific experimental cohort of cardiovascular and neurological diseases (atrial fibrillation secondary to valvular heart disease, carotid atherosclerosis, moyamoya disease)
- Healthy control group

SUMMARY:
Research purpose Using single-cell sequencing, 3D/4D genomics and multidimensional omics technologies to reveal the complex cellular and molecular regulatory networks of cardiovascular and nervous system diseases, unique phenotypic changes of specific cell types, and different gene expression patterns, identify cell types and cell subsets associated with cardiovascular and nervous system diseases, and discover disease-related genes. To reveal new pathological mechanisms of related diseases and develop new diagnosis and treatment methods.

Research background Cardiovascular and nervous system diseases such as arrhythmias (atrial fibrillation, ventricular tachycardia, ventricular fibrillation, postoperative vascular stenosis injury, etc.), heart failure, atherosclerosis (coronary heart disease, stroke, peripheral vascular disease, carotid atherosclerosis, etc.), epilepsy, moyamoya disease, etc., are currently leading to the main diseases affecting the health and death of residents in China.

The data integration method based on single-cell sequencing, multi-omics data, and machine learning to analyze molecular level changes in cardiovascular and nervous system-related diseases can help deepen the research on the pathogenesis of cardiovascular and nervous system-related diseases and provide new ideas for the prevention and treatment of related diseases.

DETAILED DESCRIPTION:
1. Test population Disease-specific experimental cohort of cardiovascular and neurological diseases (atrial fibrillation secondary to valvular heart disease, carotid atherosclerosis, moyamoya disease) and corresponding control cohort of normal tissue.
2. Sample size calculation Through literature research and clinical diagnosis experience, reliable conclusions can be obtained with an experimental cohort of 200 or more people and a control cohort. So the experimental data were selected from a disease cohort of 200 people and a control cohort of 200 people.
3. Specific research content

<!-- -->

1. Clinical data collection Clinical data (name, age, sex, weight/height ratio (BMI), three routine procedures (blood routine, stool routine, urine routine), blood biochemistry, liver and kidney function, coagulation function, bedside electrocardiogram, 24-hour holter electrocardiogram, heart color Doppler ultrasound, carotid color Doppler ultrasound, family history, past history, medication history, treatment history, and personal history) were collected from patients who met the inclusion criteria and controls Etc.), sign a written informed consent.

   1. Blood collection: Collect 5-10ml of fasting blood from the experimental population in the morning for blood routine, blood biochemistry, liver and kidney function, coagulation function and other tests.
   2. Fecal collection: 3-5g feces of the experimental population without eating from 6 a.m. to 9 a.m. will be collected for stool routine and intestinal flora detection. Note: The sample must not take antibiotics and other drugs within 45 days.
   3. Urine collection: Collect the first urine of the experimental group in the morning, and reserve 10-12ml of fresh midstream urine for routine urine detection.

      After testing the samples collected above, the test results were put into the corresponding experimental population data.
2. Single cell sequencing

   1. Sample collection and processing ① Sample collection:

      Sample collection of patients with atrial fibrillation:

      A small amount of useless left atrial appendage tissue 100mg was taken as a sample during surgical treatment of atrial fibrillation patients. (The tissue used in this study was either residual tissue or abandoned tissue, and both were necessary for surgical resection, so there was no additional risk to the subjects)

      Atrial fibrillation control heart tissue sample collection:

      Atrial fibrillation control heart tissue was 100mg of cut waste tissue from heart transplant donor heart.

      Carotid atherosclerosis sample collection:

      During the surgical treatment of carotid atherosclerotic plaque endarterectomy, at least 1mg of the central tissue of discarded vascular plaque was collected as a sample.

      Carotid atherosclerosis control sample collection:

      During the surgical treatment of carotid atherosclerotic plaque endarterectomy, at least 1mg of marginal tissue of discarded vascular plaque was collected as control samples.

      Moyamoya disease sample collection:

      During cerebrovascular bypass surgery for Moyamoya disease, at least 1mg of discarded vascular tissue was collected as a sample.

      Moyamoya disease control sample collection:

      During cerebrovascular bypass surgery in non-moyamoya disease patients, at least 1mg of pruned waste vascular tissue was collected as a sample.
      * Sample preservation and delivery: Considering that on-site experiments need to be booked in advance and coordinated, and there are many uncertain factors in clinical sample collection. For most freshly obtained samples, Miltenyi MACS Tissue Storage Solution® (130-100-008) is recommended. Optimized for the storage of fresh organ and tissue samples, the preservation solution has been tested and validated on a variety of human and mouse tissues, including tumors, skin, heart, spleen, brain, and skeletal muscle.

      Procedure for using the preservation solution: a) Collect fresh samples from the operating room or anatomy, and quickly remove non-target tissues such as fat, hair, fibers, necrotic parts, etc., within 10 minutes; b) If the tissue block is large, it is recommended to divide it into soybean size and save it or keep it for backup; c) Directly transfer the sample to the pre-cooled (2-8℃) tissue preservation solution (1.5ml EP tube) to ensure that the tissue blocks are completely covered and the sample name is well marked; d) Seal the sample tube with sealing film, separate the sample from the ice pack with foam paper, put it in a ziplock bag, and arrange the ice pack to be sent as soon as possible. a) The tissue storage solution can be stored for 48h. In order to ensure the quality of the sample, the logistics delivery should be delivered the next day or the next morning, and the mailing should be delivered in advance of the sample date. b) It is recommended to place enough ice packs to avoid complete melting, and to avoid direct contact with the sample tube, causing the sample to freeze; c) Select a foam box with a thickness of not less than 3cm, and put some ice packs into the bottom first; d) The sample tube and the ice pack should be separated by foam paper or bubble bag; It is necessary to prepare the ice pack in advance, and avoid taking the ice bag out directly from -80℃ and -20℃, otherwise the tissue block will freeze due to low temperature, resulting in tissue damage.

      ③ Digestion: Fresh heart tissue (no less than 100mg of control clipped tissue, 3-4 pieces of puncture tissue (16G puncture needle, 1.5cm)), chopped into 1~3mm3 tissue blocks, And transferred to 15 ml EP tubes of DMEM containing collagenase I (450 U ML-1), DNase I (60 U ML-1) and hyaluronidase (60 U ML-1). Incubate at 37 ° C for 1 hour, then add HBB buffer (2% FBS and 0.2% BSA in HBSS) to stop digestion, filter through a 40 µm filter into a 50 ml conical tube, transfer to a clean 15 ml EP tube and centrifuge at 4 ° C 350g for 5 min. The supernatant was then removed and the particles were re-suspended in 1 ml of ACK lysis buffer (Gibco, A10492), digested at room temperature for 5 minutes before 9 ml of DMEM was added. The supernatant was removed by centrifugation and re-suspended in 5 ml FACS buffer (2% FBS and 2mM EDTA, in a calcium/magnesium free PBS).

      ④ Sorting: Centrifugation was repeated under the above conditions, the supernatant was removed, and the cell particles were re-suspended in 300 µl cell suspension buffer (0.04%BSA, 1×PBS) and 1 µl DRAQ5 (Thermo Fisher Scientific, 62251) and 4, 6-diaminidine - 2-phenylindole (DAPI; BD Biosciences, 564907) and incubate for 5 minutes before sorting. DRAQ5+/DAPI- cells are collected in a cell re-suspension buffer. The collected cells were then re-centrifuged according to the above parameters and re-suspended in a cell re-suspension buffer to a target concentration of 1,000 cells ul-1. The cells are counted with a blood cell counter and the concentration is adjusted as needed.

      ⑤ Database building: All reagents required for database building are included in 10X Genomics Single Cell 3 'Reagent Kits v2 kit or BD database building kit.

ELIGIBILITY:
Inclusion criteria

1. Inclusion criteria for patients with valvular atrial fibrillation:

   Moderate or above mitral valve disease; The occurrence of atrial fibrillation was recorded by 12-lead electrocardiogram or 24-hour holter electrocardiogram. 3.18≤ Age ≤75 years old.
2. Inclusion criteria for disease control of valvular atrial fibrillation:

   No moderate or above mitral valve disease; No history of atrial fibrillation, 24-hour holter electrocardiogram did not record the occurrence of atrial fibrillation. 3.18≤ Age ≤75 years old.
3. Inclusion criteria for carotid atherosclerosis cases:

   Carotid atherosclerosis was confirmed by ultrasound, CTA and other imaging diagnosis. 2.18≤ Age ≤75 years old.
4. Inclusion criteria for carotid atherosclerosis control:

   The inclusion criteria for carotid atherosclerosis cases were met. The peripheral tissue of the vascular plaque was discarded in the same patient.
5. Inclusion criteria for moyamoya disease cases:

   Imaging diagnosis confirmed moyamoya disease; 2.18≤ Age ≤75 years old.
6. Moyamoya disease control inclusion criteria:

Imaging diagnosis confirmed no moyamoya disease; 2.18≤ Age ≤75 years old.

Exclusion criteria

1. Exclusion criteria for patients with valvular atrial fibrillation:

   Coronary heart disease, myocardial infarction, hyperthyroidism, severe hepatic and renal insufficiency, benign and malignant tumors, etc. Dilated cardiomyopathy, hypertrophic cardiomyopathy, congenital heart disease, heart failure and other non-valvular factors cause atrial fibrillation.
2. Exclusion criteria for control of valvular atrial fibrillation:

   Coronary heart disease, myocardial infarction, hyperthyroidism, severe hepatic and renal insufficiency, benign and malignant tumors, etc. Dilated cardiomyopathy, hypertrophic cardiomyopathy, congenital heart disease, heart failure, etc.
3. Exclusion criteria for carotid atherosclerosis cases:

   History of carotid vascular surgery or trauma
4. Exclusion criteria for carotid atherosclerosis control:

   No plaque margin tissue or marginal tissue injury was found in abandoned vessels in the same patient.
5. Exclusion criteria for moyamoya disease cases:

   Previous history of cerebrovascular surgery or trauma.
6. Exclusion criteria for moyamoya disease control:

Previous history of cerebrovascular surgery or trauma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the hospital diagnosis results, after the subjects are identified as the subjects of this experiment, they will be explained about the experiment process and informed of the benefits/risks, and they will sign the informed consent and enter the group voluntarily.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Blood collection | One month after the patient is clinically diagnosed with the above disease
  ① Collect 5-10ml blood of the subject, centrifuge, collect serum and plasma, temporarily do not test, can be immediately frozen at low temperature, the lower the temperature is better, if not repeated freezing and thawing in the middle, can be stored for one month below -20℃, can be stored for three months below -80℃.
  ② Citrate anticoagulant and plasma collection: Sodium citrate acts as an anticoagulant by acting on calcium ion chelation in blood samples, recommended by the National Committee for Standardization of Clinical Laboratories (NCCLS) is 3.2% or 3.8%, and the anticoagulant to blood ratio is 1: 9, mainly used in the fibrinolytic system (prothrombin time, thrombin time, activated partial thrombin time, fibrinogen). When taking blood, attention should be paid to taking enough blood to ensure the accuracy of the test results, and the blood should be gently reversed and mixed 5-8 times immediately after taking blood.
stool samples | One month after the patient is clinically diagnosed with the above disease
  ① Sampling should be taken at the non-eating stage between 6am and 9am Before sampling, stool must be emptied into a clean and dry urinal or container containing filter paper. Note: Urine should not be mixed into the container.
  ② Use a small spoon in the sampler to collect feces. Note: In order to prevent contamination of the stool surface, gently peel the surface with a sampling spoon, and sample the inside of the stool, placing it in an average of three feces tubes.
  ③ After sampling, close the cover of the collector and mark the name and sampling time on the collector with a pen. Store at room temperature for 1 day, long-term storage at -80℃.
  Note: The sampler should not take antibiotics or other drugs for 45 days.
urine specimen | One month after the patient is clinically diagnosed with the above disease
  The first urine of the experimental group was collected in the morning and used for urine routine detection.
  A clean, covered, disposable volume is usually used for urine collection, and the volume of the container for urine collection is generally greater than 20mL.
  The container for urine collection should be labeled, including the patient's name, the specimen code and the time of urine collection.
  Urine should be taken within two hours as soon as possible
Single cell sequencing(Disease Group) | Collected during surgical treatment
  During surgical treatment, at least 1mg of pathological waste tissue was taken as a sample The corresponding single cell samples were obtained through the steps of preservation, digestion, sorting and library building.
  Sample collection of patients with atrial fibrillation:
  A small amount of useless left atrial appendage tissue 100mg was taken as a sample during surgical treatment of atrial fibrillation patients. (The tissues used in this study were either residual tissues or abandoned tissues, and both were necessary for surgical resection, so there was no additional risk for subjects.)
  Carotid atherosclerosis samples were collected:
  During the surgical treatment of carotid atherosclerotic plaque endarterectomy, at least 1mg of the central tissue of discarded vascular plaque was collected as a sample.
  Moyamoya disease sample collection:
  During cerebrovascular bypass surgery for Moyamoya disease, at least 1mg of discarded vascular tissue was collected as a sample.
Single cell sequencing (control group) | Collected during surgical treatment
  During surgical treatment, at least 1mg of pathological waste tissue was collected as a sample .The corresponding single cell samples were obtained through the steps of preservation, digestion, sorting and library building.
  Atrial fibrillation control heart tissue sample collection:
  Atrial fibrillation control heart tissue was 100mg of cut waste tissue from heart transplant donor heart.
  Carotid atherosclerosis control sample collection:
  During the surgical treatment of carotid atherosclerotic plaque endarterectomy, at least 1mg of marginal tissue of discarded vascular plaque was collected as control samples.
  Moyamoya disease control sample collection:
  During cerebrovascular bypass surgery in non-moyamoya disease patients, at least 1mg of pruned waste vascular tissue was collected as a sample.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Tao, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Hu F, Zheng L, Liu S, Shen L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Avoidance of Vagal Response During Circumferential Pulmonary Vein Isolation: Effect of Initiating Isolation From Right Anterior Ganglionated Plexi. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007811. doi: 10.1161/CIRCEP.119.007811. Epub 2019 Nov 25. PMID 31760820
- [Background] Garnvik LE, Malmo V, Janszky I, Ellekjaer H, Wisloff U, Loennechen JP, Nes BM. Physical activity, cardiorespiratory fitness, and cardiovascular outcomes in individuals with atrial fibrillation: the HUNT study. Eur Heart J. 2020 Apr 14;41(15):1467-1475. doi: 10.1093/eurheartj/ehaa032. PMID 32047884
- [Background] Horn P, Bueltmann E, Buch CV, Schmiedek P. Arterio-embolic ischemic stroke in children with moyamoya disease. Childs Nerv Syst. 2005 Feb;21(2):104-7. doi: 10.1007/s00381-004-0962-y. Epub 2004 May 18. PMID 15148620